# Effect of Vitamin D as Adjuvant Therapy in Preterm Infants With Neonatal Sepsis

### **Informed Consent Form**

Version 1 1<sup>st</sup> June 2025

NCT Number: NCT ID not yet assigned **Unique Protocol Id:** DP. 04.03/D.XIV.6.5/337/2025

Authors: Michelle Angelica Wijaya<sup>1</sup> Reni Ghrahani<sup>1</sup> Fiva Aprilia Kadi<sup>1</sup>

Investigators:
Principal Investigator: Michelle Angelica Wijaya<sup>1</sup>
Other Investigators:
Reni Ghrahani<sup>1</sup>
Fiva Aprilia Kadi<sup>1</sup>

<sup>1</sup>Department of Child Health, Universitas Padjadjaran Medical School/Dr. Hasan Sadikin Hospital, Bandung, West Java



#### RUMAH SAKIT UMUM PUSAT Dr. HASAN SADIKIN BANDUNG

Dr. HASAN SADIKIN GENERAL HOSPITAL BANDUNG

#### **KOMITE ETIK PENELITIAN KESEHATAN**

HEALTH RESEARCH ETHICS COMMITTEE

Jl. Pasteur No. 38 Bandung 40161



Form 2

#### **INFORMATION**

"Effect of Vitamin D as Adjuvant Therapy in Preterm Infants with Neonatal Sepsis"

#### **Research Access:**

#### Research Team consists of:

| NO. | RESEARCH TEAM | PHONE |
|-----|---------------------------------------------|--------------|
| 1. | Michelle Angelica Wijaya | 081313996911 |
| 2. | Dr. Reni Ghrahani, dr., Sp.A(K)., M.Kes | 08122111482 |
| 3. | Dr. Fiva Aprilia Kadi, dr., Sp.A(K)., M.Kes | 081120050111 |

#### **Background:**

Neonatal sepsis is a disease caused by the presence of bacteria in the blood occurring in the first month of life. The immune system in infants, especially premature babies, is not fully developed, making them more susceptible to infection. Neonatal sepsis is treated by administering antibiotics via infusion. However, recent studies are still exploring various other therapies that can aid the healing process of neonatal sepsis.

Some recent research has found that vitamin D is related to sepsis. Vitamin D plays a role in the immune system and can help accelerate the reduction of inflammation markers and infection in the body. Vitamin D also has a low risk of toxicity/overdose, minimal side effects, and is affordable. Research on the effect of vitamin D as an adjuvant therapy in neonatal sepsis is still very limited globally, and in Indonesia, there have been no similar studies to date.

#### **Objective:**

To evaluate the effect of vitamin D administration as an adjuvant therapy in neonatal sepsis by measuring differences in sepsis scores and CRP levels.

#### Why your child is selected:

Your child meets the criteria, which is being a premature infant diagnosed with neonatal sepsis and without any major congenital abnormalities.

#### **Benefits:**

Your child's vitamin D levels will be examined and, if possible (if able to take orally), will be given additional vitamin D therapy. It is hoped that by understanding the effect of vitamin D as an adjunct therapy for neonatal sepsis, it can serve as a consideration for vitamin D administration in such cases.

#### **Potential Discomfort and Risks:**

Pain during blood sampling: Pain management for infants will be provided, such as pacifiers with sugar/breastmilk. Risk of infection and bruising/hematoma: Sterile equipment will be used, and antiseptic techniques applied before

blood collection. Bruises will be treated with a cold compress using gauze and 0.9% NaCl infusion fluid.

#### Possibility of Unknown Risks:

Vitamin D overdose/toxicity, such as excess calcium levels in the blood.

#### **Procedure:**

- Parents/guardians of participants diagnosed with neonatal sepsis and who meet the research criteria will be given a detailed explanation of the research, and after agreeing, will be asked to sign an informed consent form.
- 2. Blood samples of 4 mL will be taken from a vein on Day 0 and Day 7, along with other evaluation blood tests.
- 3. Patients selected for the treatment group will receive additional vitamin D3 (either 1x400 IU or 1x800 IU daily) for 7 days, with laboratory evaluation done on Day 0 and Day 7.
- 4. Data will be collected and statistically analyzed.

#### **Complications and Compensation:**

Medical treatment will be provided if there's any complication related to this study

#### Can the subjects be withdrawn or withdraw themselves from the study?:

Yes

#### **Data Confidentiality:**

Your child's data will be kept confidential

Bandung, 1<sup>st</sup> June 2025 Principal Investigator

Michelle Angelica Wijaya



## INFORMED CONSENT FORM TO PARTICIPATE IN RESEARCH

Jl. Pasteur No. 38 Bandung

#### INFORMATION

Principal Investigator: dr. Michelle Angelica Wijaya

Name of the person providing information:

Research participant:

Witness:

| NO | INFORMATION | CONTENT O | OF INFORMATION |
|---|---|---|---|
| 1 | Explanation about the research, duration of the research subject's participation, and procedures that must be followed by the subject | The study will be conducted for 7 days from the time the patient is diagnosed with neonatal sepsis. Blood samples will be taken twice, on day 0 and day 7, with a volume of 4 mL each time. For patients who are not fasting, those in the treatment group will be given additional vitamin D3 at a dose of 1x400 IU (0.5 mL) or 1x800 IU (1 mL) daily for 7 days, in addition to antibiotic administration. | |
| 2 | Expected benefits | Subjects participating in the study can know their 25(OH)D levels, and those in the treatment group will receive vitamin D3 supplementation as an additional therapy. | |
| 3 | Potential discomforts and risks that may arise | Pain during blood collection | |
| 4 | Alternative treatments and procedures that also provide benefits | None | |
| 5 | Maintain the confidentiality of research data | The confidentiality of the subject's data is guaranteed. | |
| 6 | Provision of compensation or medical treatment if complications occur | Yes, medical treatment will be provided | |
| 7 | Participation is voluntary | Participation in this research is voluntary. | |
| 8 | Refusal to participate or withdrawal from the study will not affect your access to hospital services, nor will it compromise the care you receive. | The parent/guardian of the subject has the right to refuse participation and will not face any penalties, nor will it compromise the care or access to hospital services. | |
| 9 | If you have any questions or need more information, please contact | Michelle (Phone: 081313996911) | |
| 10 | Others | None | |
| | by declare that I (principal investigator) have explain | | Principal Investigator |
| | rs correctly and clearly, and have provided the oppoions and/or discuss. | riunity to ask | (Michelle Angelica) |

| I hereby declare that I (the patient's guardian) have received the information | Patient's guardian*) |
|---|---|
| from the person in charge of the research as stated above and have | |
| understood it. | |
| | () |
| | Signature and name |
| | Witness |
| | () |
| | Signature and name |

RM.IC.06/15

#### STATEMENT OF CONSENT

| The person(s) signing below: | | |
|---|---|---|
| Medical record : | | |
| "Effect of Vitamin D as Adjuvant Therapy in Preterm Infants with Neonatal Sepsis" | | |
| herefore, I declare: Agree / Disagree*) to let my child participate in this research. This statement is made truthfully and without any coercion, | | |
| Bandung, | | |
| The undersigned. | Principal Investigator | Witness |
| () Signature and name | (dr. Michelle Angelica Wijaya)<br>Signature and name | () Signature and name |

RM.IC.06/15



#### RUMAH SAKIT UMUM PUSAT Dr. HASAN SADIKIN BANDUNG

Dr. HASAN SADIKIN GENERAL HOSPITAL BANDUNG

#### **KOMITE ETIK PENELITIAN KESEHATAN**







Form 3

#### STATEMENT OF CONSENT TO PARTICIPATE IN RESEARCH (INFORMED CONSENT)

| The undersigned: | | | | |
|---|---|---|---|---|
| Name: | | | | |
| Age: | | | | |
| Address: | | | | |
| Occupation: | | | | |
| ID Number: | | | | |
| Who is the parent/guard | dian of: | | | |
| Name | : | | | |
| Medical Record | : | | | |
| Age | : | | | |
| Address | : | | | |
| Hereby declare that: | | | | |
| | explanation, I am fully aware o<br>y arise in this research, and that | | | • |
| "Effect of Vitamin D a | as Adjuvant Therapy in Pretern | n Infants with Neonata | al Sepsis" | |
| Therefore, I hereby decla <b>Agree and give permissi</b> | re:<br>ion / Do not agree and do not | give permission* for n | ny child to parti | cipate in this research. |
| This statement is made tr | uthfully and without coercion. | | | |
| Witnesses: | | Bandur | ng, | 2025 |
| | | Parent/ | guardian of the | research participant |
| () | | | | |
| | | ( | | , |
| | | ( | | <i>)</i> |
| () | | | | |

(\*) The participant can select either "Agree and give permission" or "Do not agree and do not give permission."